CLINICAL TRIAL: NCT00003768
Title: A Phase I Pharmacokinetic Study of Single Dose Intravenous CA4P in Patients With Advanced Cancer
Brief Title: Combretastatin A4 Phosphate in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILEX1Y98; CWRU-ILEX-1Y98; ILEX-1Y98; ILEX-CA4P101-A3; NCI-G99-1502
Record Dates: First submitted 2000-04-06; First posted 2004-05-03 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — fosbretabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fosbretabulin disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of combretastatin A4 phosphate in treating patients who have advanced solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of combretastatin A4 phosphate when administered at single doses every 21 days in patients with advanced solid tumors. II. Determine both the toxicity and dose limiting toxicity of this regimen in these patients. III. Determine the plasma and urine pharmacokinetics of combretastatin A4 and combretastatin A4 phosphate. IV. Gather preliminary data regarding possible antitumor effects in those patients with measurable disease.

OUTLINE: This is an open label, dose escalation study. Patients receive combretastatin A4 phosphate IV over 10-60 minutes. Treatment repeats every 3 weeks in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of combretastatin A4 phosphate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity. Patients are followed at 3 weeks.

PROJECTED ACCRUAL: A maximum of 21 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven advanced solid tumors that have failed standard therapy or for which no curative therapy exists No leukemia, lymphoma, or multiple myeloma No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin normal SGOT/SGPT no greater than 3 times upper limit of normal (ULN) PT/PTT less than ULN OR International normalized ratio (INR) less than 1.1 Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No clear evidence of acute ischemic heart disease on EKG No history of myocardial infarction within past 6 months No history of angina No peripheral vascular disorder Neurologic: No active seizure disorder Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No evidence of hematemesis, melena, or hematochezia No history of inflammatory bowel disease, autoimmune disease, or bleeding disorders No Type I diabetes mellitus or Type II diabetes with peripheral vascular disorders No active infections or any serious concurrent systemic disorders incompatible with study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosoureas) and recovered No other concurrent cytotoxic therapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: At least 6 weeks since prior major surgery Other: At least 4 weeks since any other prior investigational agent No concurrent anticonvulsant therapy No concurrent aspirin greater than 100 mg per day, heparin, or nonsteroidal antiinflammatory medication No concurrent calcium channel blockers, antiarrhythmias, or anti-angina therapy Concurrent beta-blocking agents for hypertension or anxiety allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1998-09; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Giri P, Batra PJ, Kumari A, Hura N, Adhikary R, Acharya A, Guchhait SK, Panda D. Development of QTMP: A promising anticancer agent through NP-Privileged Motif-Driven structural modulation. Bioorg Med Chem. 2023 Nov 15;95:117489. doi: 10.1016/j.bmc.2023.117489. Epub 2023 Oct 5. PMID 37816266